CLINICAL TRIAL: NCT06459973
Title: A Multi-center, Open-label, Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of YL205 in Patients With Advanced Solid Tumors
Brief Title: A Clinical Study of YL205 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YL205-CN-101-01
Record Dates: First submitted 2024-05-30; First posted 2024-06-14 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase Ia: Dose escalation portion (Experimental): YL205 is provided as the lyophilized powder, 160 mg/vial. Adcanced solid tumors patients will be given YL205 by intravenously once every 3 weeks (Q3W) as a cycle at several dose levels.
  Interventions: Drug: intravenous (IV) infusion
- Phase Ib: Dose expansion portion (Experimental): YL205 is provided as the lyophilized powder, 160 mg/vial. Adcanced solid tumors patients will be given YL205 by intravenously once every 3 weeks (Q3W) as a cycle at no less than two dose levels.
  Interventions: Drug: intravenous (IV) infusion
- Phase II: Cohort expansion portion (Experimental): YL205 is provided as the lyophilized powder, 160 mg/vial. Adcanced solid tumors patients will be given YL205 by intravenously once every 3 weeks (Q3W) as a cycle at RP2D.
  Interventions: Drug: intravenous (IV) infusion

INTERVENTIONS:
Drug: intravenous (IV) infusion — YL205 is provided in the form of lyophilized powder under a strength of 160 mg/vial. Each vial should be reconstituted to 20 mg/mL. Prior to IV infusionSubjects will be treated with YL205 via intravenous (IV) infusion, once every 3 weeks (Q3W) as a treatment cycle

SUMMARY:
This study is a multicenter, open-label, phase I/II study of YL205 in China to evaluate the safety, tolerability, PK characteristics and preliminary efficacy of YL205 in the following selected patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subjects who are informed of relevant information of the study prior to initiation of the study and voluntarily sign and date on the informed consent form (ICF).

  2) Age ≥18 years. 3) Be willing to follow and be able to complete all the study procedures. 4) Body mass index (BMI) within the range of 18 to 32 kg/m2, and body weight ≥45kg for female subjects.

  5） Patients with histologically or cytologically confirmed locally advanced or metastatic ovarian cancer (OC), non-squamous non-small cell lung cancer (NSQ NSCLC), renal cell carcinoma (RCC), endometrial cancer (EC), or other Napi2b-overexpressing tumors。 6) Patients with positive Napi2b test results at the central laboratory. 9) At least one radiologically evaluable lesion for subjects in Part 1; At least one measurable extracranial lesion (non-radiation fields) for subjects in Part 2 and Part 3.

  10) Expected survival ≥3 months. 11) Female subjects of childbearing potential must agree to take effective contraceptive measures and must not undergo egg donation or egg retrieval for their own use from screening throughout the study period and for at least 6 months after the last dose of the investigational drug. Male subjects must agree to take effective contraceptive measures and must not undergo sperm cryopreservation or sperm donation from screening throughout the study period and for at least 6 months after the last dose of the investigational drug.

  12) subjects must provide tumor samples. 13) Subjects who are capable of and willing to comply with the visits and procedures stipulated in the study protocol.

Exclusion Criteria:

* 1) Subjects with a treatment history with drugs targeting Napi2b. 2) Subjects with a history of intolerance to topoisomerase I inhibitors or ADC therapy.

  3) Subjects who are participating in another clinical study, with the exception an of observational (non-interventional) clinical study or the follow-up period of an interventional study.

  4) Subjects with an insufficient washout period from the previous anti-tumor therapy to the first dose.

  5) Subjects who received radiotherapy, including palliative stereotactic radiotherapy on the abdomen, within 4 weeks prior to the first dose.

  6) Subjects who received major surgery within 4 weeks prior to the first dose or those who plan to receive major surgery during the study.

  7) Subjects who received allogeneic bone marrow transplantation or solid organ transplantation.

  8) Subjects who received systemic steroids or other immunosuppressive treatment within 2 weeks prior to the first dose of the investigational drug.

  9) Subjects who received any live vaccine within 4 weeks prior to the first dose or those who plan to receive live vaccines during the study.

  10) Subjects with a medical history of leptomeningeal carcinoma or cancerous meningitis.

  11) Subjects with brain metastasis or spinal cord compression. 12) Subjects with uncontrolled or clinically significant cardiovascular and cerebrovascular diseases.

  13) Subjects who were diagnosed with Gilbert's syndrome. 14) Subjects with significantly symptomatic or unstable effusion in the third space requiring repeated drainage.

  15) Subjects with medical history of gastrointestinal perforation and/or fistula within 6 months prior to the first dose, or active gastric ulcers, duodenal ulcer, colitis ulcerative, or other gastrointestinal disorders that may cause hemorrhage or perforation in the opinion of the investigator.

  16) Subjects with serious infection (Grade ≥3 as per NCI CTCAE v5.0) prior to the first dose.

  17) Subjects with human immunodeficiency virus (HIV), active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection; subjects with positive syphilis antibody and a positive titer result.

  18) Subjects with unresolved toxicity caused by previous anti-tumor therapy. 20) Subjects with a history of serious allergic reactions to drugs, inactive ingredients in drug products, or other monoclonal antibodies.

  21) Female subjects who are pregnant as confirmed by a pregnancy test within 3 days prior to the first dose, or lactating women.

  22) Subjects who have any diseases, medical conditions, organ system dysfunction, or social conditions.

  23) Subjects with multiple primary malignancies within 5 years prior to the signing of the ICF, except for fully resected non-melanoma skin cancer, radically treated carcinoma in situ, or other radically treated solid tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
To evalue the DLTs | Approximately within 36 months
To evalue the TEAEs | Approximately within 36 months
  Treatment Emergent Adverse Event
To evalue the TRAEs | Approximately within 36 months
  Treatment Related Adverse Event
To evalue the serious adverse events (SAEs) | Approximately within 36 months
Determination of the MTD of YL205 in the pivotal clinical study | Approximately within 36 months
Determination of the RED of YL205 in the pivotal clinical study | Approximately within 36 months
Determination of the RP2D of YL205 in the pivotal clinical study | Approximately within 36 months
Assessed ORR (the proportion of CR and PR) by the investigator per RECIST v1.1 | Approximately within 36 months

SECONDARY OUTCOMES:
Characterize the PK parameter AUC | Approximately within 36 months
  area under curve (AUC)
Characterize the PK parameter Cmax | Approximately within 36 months
  maximum concentration (Cmax)
Characterize the PK parameter Ctrough | Approximately within 36 months
  minimum concentration at trough (Ctrough)
Characterize the PK parameter Vd | Approximately within 36 months
  volume of distribution (Vd)
Characterize the PK parameter CL | Approximately within 36 months
  plasma clearance (CL)
Characterize the PK parameter Tmax | Approximately within 36 months
  time to maximum concentration (Tmax)
Characterize the PK parameter t1/2 | Approximately within 36 months
  half-life (t1/2)
Assessed the disease control rate (DCR) per RECIST v1.1 | Approximately within 36 months
  (defined as the proportion of CR, PR, or stable disease (SD))
Assessed the duration of response (DOR) per RECIST v1.1 | Approximately within 36 months
Assessed the time to response (TTR) per RECIST v1.1 | Approximately within 36 months
Assessed the progression free survival (PFS) per RECIST v1.1 | Approximately within 36 months
Assessed the depth of response (DpR) per RECIST v1.1 | Approximately within 36 months
  the percentage change in target lesion size
Assessed the overall survival (OS) per RECIST v1.1 | Approximately within 36 months
Evaluate the corelaton between different levels of Napi2B expression and the sum of CR rate, PR rate and SD rate | Approximately within 36 months

CONTACTS AND LOCATIONS:
Locations (43):
- United States (11):
  - Sarah Cannon Research Institute (SCRI)- Denver, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists - Lake Mary, Lake Mary, Florida
  - Norton Cancer Institute, Louisville, Kentucky
  - Washington University School of Medicine - Center for advanced Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada (CCCN) - Central Valley, Las Vegas, Nevada
  - Southwest Women's Oncology, Albuquerque, New Mexico
  - Stephenson Cancer Center (Oklahoma), Oklahoma City, Oklahoma
  - Providence Cancer Institute - Franz Clinic, Portland, Oregon
  - Sarah Cannon Research (SCRI)-Tennessee, Nashville, Texas
  - University of Washington, Seattle, Washington
- China (32):
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-Sen Memorial Hospital,Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jingzhou First People's Hospital, Jingzhou, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Medical College of Hust TongJi Hospital, Wuhan, Hubei
  - Union hospital Tongji Medical Colllege Huazhong University of School and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Provincial Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jilin Provincial Cancer Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of XI'AN Jiaotong University, Xi’an, Shanxi
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital. Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - Chinese People's Liberation Army Army Characterstic Medical Center, Chongqing
  - Chongqing Cancer Hospital, Chongqing
  - The Southwest Hospital of AMU, Chongqing
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai